CLINICAL TRIAL: NCT05367700
Title: A Phase I, Open-label, Multicenter Study to Evaluate Safety, Tolerability, Pharmacokinetics, and Efficacy of Single and Multiple Doses of Oral Administration of HS-10382 in Patients With Chronic Myeloid Leukemia.
Brief Title: A Study of HS-10382 in Patients With Chronic Myeloid Leukemia.
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: Jiangsu Hansoh Pharmaceutical Co., Ltd. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Treatment
Other Study IDs: HS-10382-101
Record Dates: First submitted 2022-05-06; First posted 2022-05-10 (Actual); Last update posted 2023-01-13 (Actual); Status verified 2023-01

CONDITIONS: CML, Chronic Phase; CML, Accelerated Phase
Keywords: CML-CP/AP; HS-10382; BCR-ABL TKI; Phase I; Allosteric inhibitor
MeSH Terms: conditions — Leukemia, Myeloid, Chronic-Phase; Leukemia, Myeloid, Accelerated Phase

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- HS-10382 (Part 1: Dose escalation) (Experimental): There are five escalation dose cohorts.
  Interventions: Drug: HS-10382(Part 1: Dose escalation)
- HS-10382 (Part 2: Dose expansion) (Experimental): The recommended dose from the dose-escalation stage and other potential doses will be further explored.
  Interventions: Drug: HS-10382(Part 2: Dose expansion)

INTERVENTIONS:
Drug: HS-10382(Part 1: Dose escalation) — Single or multiple dose(s) of HS-10382 once daily.
  Arms: HS-10382 (Part 1: Dose escalation)
Drug: HS-10382(Part 2: Dose expansion) — HS-10382 is administered orally once daily.
  Arms: HS-10382 (Part 2: Dose expansion)

SUMMARY:
HS-10382 is a small molecular, oral potent, allosteric inhibitor. By binding a myristoyl site of the BCR-ABL1 protein, HS-10382 locks BCR-ABL1 into an inactive conformation. The purpose of this study is to investigate the safety/tolerability and the pharmacokinetic(PK) profile of HS-10382 in patients with chronic myeloid leukemia (CML). Anti-CML activity will also be investigated in this study.

DETAILED DESCRIPTION:
This is an open-label, multicenter, dose-escalation and expansion, first-in-human study in participants of CML with T315I mutation or without T315I mutation in chronic phase/accelerate phase(CP/AP). This study will consist of two parts: A part 1 dose escalation stage and a part 2 dose expansion stage. The objectives of this study are to evaluate the safety, tolerability, PK and preliminary anti-CML activity, describe the dose-limiting toxicities (DLTs), and determine the maximum tolerated dose (MTD) or maximum applicable dose (MAD) of HS-10382. Participants with CML-CP/AP are eligible for dose escalation study if they had resistance to or unacceptable side effect from BCR-ABL1 TKIs. After determination of the MTD or the MAD for CML patients, dose expansion will be undertaken to further evaluate the efficacy and safety of HS-10382 in patients with CML-CP. All patients will be carefully followed for adverse events during the study treatment and for 28 days after the last dose of study drug. Subjects of this study will be permitted to continue therapy with assessments for progression if the product is well tolerated and the subject has stable disease or better.

ELIGIBILITY:
Inclusion Criteria:

1. Signed informed consent form.
2. Men or women aged more than or equal to (≥) 18 years, and less than (<) 75 years.
3. CML-CP/AP patients with the Ph chromosome or BCR-ABL1 fusion genes.
4. Patient with CML-CP/AP who are resistant to or intolerant to previous TKIs therapy.
5. ECOG performance status of 0-2.
6. Life expectancy ≥ 12 weeks.
7. Men or women should be using adequate contraceptive measures throughout the study; Females should not be breastfeeding at the time of screening, during the study and until 6 months after completion of the study.
8. Females must have evidence of non-childbearing potential.

Exclusion Criteria:

1. CML-CP patients who have acquired CCyR and have not lost it.
2. Patients with CML-CP who have progressed to AP or blast phase(BP.)
3. Patients with CML-AP who have obtained CHR or no evidence of CML in peripheral blood.
4. Patients with CML-AP who have progressed to BP.
5. Previous treatment with a BCR-ABL1 TKI allosteric inhibitor .
6. Impaired cardiac function including any one of the following:

   1. Resting corrected QT interval (QTc) > 470 ms obtained from electrocardiogram (ECG), using the screening clinic's ECG machine and Fridericia's formula for QT interval correction (QTcF).
   2. Any clinically important abnormalities in rhythm, conduction, or morphology of the resting ECG.
   3. Any factors that increase the risk of QTc prolongation or risk of arrhythmic events,
   4. Left ventricular ejection fraction (LVEF) ≤ 50%.
   5. During screening period, ECG examination showed average heart rate <50 beats per minute.
   6. Myocardial infarction occurred within 6 months of the first scheduled dose of HS-10382.;
   7. Congestive heart failure occurred within 6 months of the first scheduled dose of HS-10382.;
   8. Uncontrollable angina.
7. History of acute pancreatitis within 1 year of study entry or past medical history of chronic pancreatitis
8. Any severe or uncontrolled systemic diseases (i.e. uncontrolled hypertension or diabetes).
9. Clinically severe gastrointestinal dysfunction that may affect drug intake, transport or absorption.
10. Severe infection within 4 weeks prior to the first scheduled dose of HS-10382.
11. History of significant congenital or acquired bleeding disorders unrelated to CML.
12. Inadequate other organ function.
13. History of other malignancies.
14. History of hypersensitivity to any active or inactive ingredient of HS-10382.
15. History of neuropathy or mental disorders, including epilepsy and dementia.
16. Judgment by the investigator that the patient should not participate in the study if the patient is unlikely to comply with study procedures, restrictions, and requirements.

Ages: 18 Years to 74 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 108 (Estimated)
Dates: Start 2022-04-28 (Actual); Primary Completion 2024-12-30 (Estimated); Study Completion 2026-09-30 (Estimated)

PRIMARY OUTCOMES:
Part 1(Dose escalation): Maximum tolerated dose (MTD) for HS-10382 | From the single dose to the last dose of the first cycle as 28days of multiple dosing (35days).
  MTD was defined as the previous dose level at which 2 out of 3 subjects or 2 out of 6 subjects experienced a DLT.
Part 2(Dose expansion): Major cytogenetic response (MCyR) rate at 6 months | 6 months
  MCyR is the proportion of patients achieving Complete cytogenetic response (CCyR: defined as 0% Philadelphia chromosome-positive [Ph+] metaphases by cytogenetic analysis of bone marrow) and Partial Cytogenetic Response (PCyR: defined as >0% to 35% Ph+ metaphases by cytogenetic analysis of bone marrow).

SECONDARY OUTCOMES:
Incidence and severity of treatment-emergent adverse events | From baseline until 28 days after the last dose.
  Assessed by number and severity of adverse events as recorded on the case report form, vital signs, laboratory variables, physical examination, electrocardiogram, and NCI CTCAE v5.0.
Observed maximum plasma concentration (Cmax) after single dose of HS-10382 | In the study of single-dose, Cmax will be obtained following administration of a single oral dose of HS-10382 on Day 1 to Day 6.
  From pre-dose to 120 hours after single dose on Day 1
Time to reach maximum plasma concentration (Tmax) after single dose of HS-10382 | From pre-dose to 120 hours after single dose on Day 1
  In the study of single-dose, Tmax will be obtained following administration of a single oral dose of HS-10382 on Day 1 to Day 6.
Area under plasma concentration versus time curve from zero to last sampling time (AUC0-t) after single dose of HS-10382 | From pre-dose to 120 hours after single dose on Day 1
  Area under the plasma concentration versus time curve from time zero to the last sampling time t at which the concentration was at or above the lower limit of quantification (LLQ). AUC0-t was to be calculated according to the mixed log-linear trapezoidal rule.
Hematologic response | at screening and 28th day of cycle 1,2,3,4,5,6,9 and 12.
  Hematologic response will be assessed by complete blood count (CBC) and physical examination at each visit.
Molecular response | at screening and 28th day of cycle 3, 6, 9 and 12.
  Molecular response will be assessed by BCR-ABL1 transcript level as measured by RQ-PCR.
Cytogenetic response | at screening and 28th day of cycle 3, 6, 9 and 12.
  Cytogenetic response (CyR) is based on the prevalence of Ph+ cells in metaphase from bone marrow (BM) sample.
Event-free survival (EFS) | up to 24 months
  EFS is defined as the time from the date of first dose to the earliest occurrence of the following events: death due to any cause ; loss of CHR ,loss of PCyR ;loss of CCyR ; discontinuation of study treatment due to AE or treatment failure ; progression to AP/BC .
Progression-free survival (PFS) | up to 24 months
  PFS is defined as the time from the date of first dose to the earliest occurrence of progression to AP/BC or death from any cause.
Overall survival (OS) | up to 24 months
  OS is defined as the time from the date of first dose to the date of death from any cause.

CONTACTS AND LOCATIONS:
Overall Officials: Yu Hu, Principal Investigator — Union Hospital, Tongji Medical College, Huazhong University of Science and Technology
Locations (1):
- Union Hospital affiliated to Tongji Medical College of Huazhong University of Science and Technology, Wuhan, Hubei, China